CLINICAL TRIAL: NCT02841202
Title: The Effect of Oral Contraceptive Pills On Macula, Retinal Nerve Fiber Layer and Choroid Thickness
Brief Title: The Effect of Oral Contraceptive Pills On Eyes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf MADENDAG, obstetrics and gynecology, Kayseri Education and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2013/65
Record Dates: First submitted 2016-07-14; First posted 2016-07-22 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2016-07

CONDITIONS: Adverse Effect of Oral Contraceptives, Subsequent Encounter
Keywords: optical coherence tomography; oral contraceptive pills
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- oral contraceptive pills group (Active Comparator): healthy women using oral contraceptive pills for only contraception for more than one year was called OCP group
  Interventions: Drug: oral contraceptive pills
- control group (No Intervention): The second group was called control group consisting 20 healthy women and using no drug

INTERVENTIONS:
Drug: oral contraceptive pills
  Other Names: yasmin
  Arms: oral contraceptive pills group

SUMMARY:
The investigators aimed to evaluate the effect of oral contraceptive pills(OCP) on macula, retinal nerve fiber layer and choroid thickness by using Optical Coherence Tomography (OCT). The present clinical study is the first research reported in the literature which is investigating the posterior ocular segment changes in women using OCP by using OCT.

DETAILED DESCRIPTION:
Spectral-domain optical coherence tomography (OCT) which is used to evaluate retina both qualitatively and qualitatively is a non invasive process. And also OCT makes it possible to perform retinal exams repeatedly without eye drops and dilatation.

ELIGIBILITY:
Inclusion Criteria:

* All the participants in the study group were Caucasian origin and the ages of them ranged from 18 to 48 in the reproductive period

Exclusion Criteria:

* None of the women in the study was pregnant. Women who reported histories of any medical problems such as thyroid disorders, hypertension, thromboembolic disease, diabetes mellitus, cardiovascular events, Cushing disease, positive malignancy, congenital adrenal hyperplasia, liver disease, psychotic disorders and neither did they use antidepressants nor steroidal hormone drugs and mood stabilizers (lithium, valproic acid, cocaine, antiandrogens, and insulin sensitizers, etc) were excluded from the study. Subjects were also excluded if they used caffeine or tobacco. The investigators also excluded from the study those women who had ocular surgery, ocular trauma or any ocular diseases such as glaucoma, cystoid macular edema, macular degeneration, optic atrophy, intraocular pressure 421 mmHg, cataract, best corrected visual acuity worse than 20/30, high spherical4± 3 dioptre or cylindrical42 dioptre refractive errors and uveitis at the time of OCT measurement.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events on Eyes That Are Related to Treatment | one year

CONTACTS AND LOCATIONS:
Overall Officials: YUSUF MADENDAG, Principal Investigator — Kayseri Education and Research Hospital